CLINICAL TRIAL: NCT03611387
Title: Artificial Intelligence Screening on Patients With Primary Angle Closure Glaucoma
Acronym: AI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: University of California (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Sun Yat-sen University
Other Study IDs: CCPMOH2018-China-4
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Ophthalmopathy
Keywords: Primary Angle-Closure Glaucoma; Artificial Intelligence
MeSH Terms: conditions — Eye Diseases; Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal: Patients without any type of glaucoma
  Interventions: Device: CASIA 2 OCT
- Primary angle closure glaucoma: Patients with primary angle closure glaucoma
  Interventions: Device: CASIA 2 OCT
- Primary open-angle glaucoma: Patients with primary open-angle glaucoma
  Interventions: Device: CASIA 2 OCT

INTERVENTIONS:
Device: CASIA 2 OCT — Using CASIA 2 OCT to assess the anterior chamber angle of the eye in the glaucomatous patients withconventional imaging methods

SUMMARY:
The Tomey CASIA (Tomey Corporation, Nagoya, Japan) is a novel rapid imaging device that captures high-quality imaging of the entire anterior chamber of the eye over detailed imaging of a single section. In this prospective study, we want to investigate and compare the anatomical structure of the drainage angle of the eye in patients with different types glaucoma using Tomey machine. This study gives us a better understanding of the predictability, validity and accuracy of Tomey machine in the diagnosis of different types of glaucoma. Moreover, the data collected here will be used to create an artificial intelligence (AI) platform to screen certain type of glaucoma.

DETAILED DESCRIPTION:
Patients ≥18 years old from ophthalmic clinics with or without glaucoma were enrolled to this respective observational clinical study. However, patients with any history of eye surgery (except cataract surgery) including laser procedure were excluded. The investigators will review patients' medical chart and update any medical history in your medical record. If new scans are needed, investigators will do them at the time of patients' current visit and it will require about 30 mins. CASIA SS-OCT (CASIA 2) is a non-contact scan of the front of the eye with higher resolution and provides deeper, wider and three- dimensional views. It is the newest scan machine. It is not FDA-approved but is approved in many other countries including Japan for patient use. We may perform the scan in the light and dark condition. We may also perform the routine scan to capture images of the anterior part of the eye for comparison purpose. The results of the scanned data will be among patients' medical records. Age, sex and ethnicity within your medical records will also be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with or without glaucoma

Exclusion Criteria:

* Patients with any history of eye surgery (except cataract surgery) including laser procedure.
* Age < =18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients ≥18 years old with or without glaucoma
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The accuracy of the CASIA 2 OCT | baseline
  To compare the clinical applicability, accuracy, and validity of the CASIA 2 OCT (Tomey, Nagoya, Japan) in the assessment of anterior chamber angle of the eye in the glaucomatous patients withconventional imaging methods.
The sensitivity and specificity of the AI | baseline
  To create an AI program to reliably screen patients with certain type of glaucoma (such as primary angle closure glaucoma, PACG) using images from CASIA 2 OCT. To test the sensitivity and specificity of the AI program to screen patients with glaucoma using images from CASIA 2 OCT. Another database comprised of CASIA 2 OCT images will be created and used to test the AI program. The diagnosis based on the AI program will be compared with diagnosis from glaucoma specialist.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China